CLINICAL TRIAL: NCT05913076
Title: Evaluation of the Effects of Alternating Rapid Maxillary Expansion and Facemask Use in Cases of Class III Malocclusion Caused by Maxillary Retrognathia- A Prospective, Randomized Clinical Trial
Brief Title: Class III Malocclusion and ALT-RAMEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Hande Uzunçıbuk, Research Assistant Dr./ Principal Investigator, Trakya University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: facemasktrakya1234
Record Dates: First submitted 2023-05-17; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Face Mask; Rapid Maxillary Expansion; Maxillary Retrognathism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigation of the Effects of Alt-RAMEC and Facemask 1 week Use in Class III Malocclusion (Experimental): A sample of 40 patients, consisting of 18 males and 22 females with a mean age of 10.64 ± 0.98, who were in the growth and developmental stage, were divided into three treatment groups. The formation of groups was carried out with the aim of achieving a near-equal distribution of male and female participants within each group, as indicated in Table 1. The first group comprised 14 patients, while the second and third groups consisted of 13 patients each. The skeletal age of the individual was determined through the acquisition of hand-wrist X-rays and the application of the Greulich and Pyle atlas at T1.
  Interventions: Device: Delaire Face Mask (M0774-01, Leone S.p.A., Florence, Italy) for first group
- Investigation of the Effects of Alt-RAMEC and Facemask 3 week Use in Class III Malocclusion (Experimental): The second group comprised 13 patients who were in the growth and developmental stage. The skeletal age of the individual was determined through the acquisition of hand-wrist X-rays and the application of the Greulich and Pyle atlas at T1.
  Interventions: Device: Delaire Face Mask (M0774-01, Leone S.p.A., Florence, Italy) for second group
- Investigation of the Effects of Alt-RAMEC and Facemask 5 week Use in Class III Malocclusion (Experimental): The third group comprised 13 patients who were in the growth and developmental stage. The skeletal age of the individual was determined through the acquisition of hand-wrist X-rays and the application of the Greulich and Pyle atlas at T1.
  Interventions: Device: Delaire Face Mask (M0774-01, Leone S.p.A., Florence, Italy) for third group

INTERVENTIONS:
Device: Delaire Face Mask (M0774-01, Leone S.p.A., Florence, Italy) for first group — The study involved the fabrication of occlusal-coverage bonded type RME devices utilizing Hyrax screws (A0620-11, Leone S.p.A., Firenze, Italy). Each patient in Group 1 (classical RME method) was instructed to open Hyrax screw twice a day for a week. At the end of the respective periods (1 week), the screws were fixed with ligatures, and the patients were evaluated.
  Face-mask treatment was subsequently started after RME. Totaling 700 g of extraoral traction force applied to maxilla. Patients were advised to wear Delaire type facemasks (M0774-00, Leone SpA) 14-16 hours a day for 6 months.
  Other Names: (Fabricated for every patient) Bonded-type Expansion Device
  Arms: Investigation of the Effects of Alt-RAMEC and Facemask 1 week Use in Class III Malocclusion
Device: Delaire Face Mask (M0774-01, Leone S.p.A., Florence, Italy) for second group — The same fabrication of occlusal-coverage bonded type RME devices were utilized Hyrax screws (A0620-11, Leone S.p.A., Firenze, Italy) in Group 2. Each patient in Group 2 (3-week Alt-RAMEC protocol), the patients were instructed to activate Hyrax screw twice a day for one week, close the screw for following week, and open the screw over the third week. At the end of the respective periods (3 weeks), the screws were fixed with ligatures, and the patients were evaluated.
  Face-mask treatment was subsequently started after RME. Totaling 700 g of extraoral traction force applied to maxilla. Patients were advised to wear Delaire type facemasks (M0774-00, Leone SpA) 14-16 hours a day for 6 months.
  Other Names: (Fabricated for every patient) Bonded-type Expansion Device
  Arms: Investigation of the Effects of Alt-RAMEC and Facemask 3 week Use in Class III Malocclusion
Device: Delaire Face Mask (M0774-01, Leone S.p.A., Florence, Italy) for third group — The same fabrication of occlusal-coverage bonded type RME devices were utilized Hyrax screws (A0620-11, Leone S.p.A., Firenze, Italy) in Group 3. Each patient in Group 3 (5-week Alt-RAMEC protocol), the patients were instructed to activate Hyrax screw twice a day for one week, close the screw for following week, and open the screw over the third week. The aforementioned screw open-close procedure was implemented over a period of five weeks. At the end of the respective periods (5 weeks), the screws were fixed with ligatures, and the patients were evaluated.
  Face-mask treatment was subsequently started after RME. Totaling 700 g of extraoral traction force applied to maxilla. Patients were advised to wear Delaire type facemasks (M0774-00, Leone SpA) 14-16 hours a day for 6 months.
  Other Names: (Fabricated for every patient) Bonded-type Expansion Device
  Arms: Investigation of the Effects of Alt-RAMEC and Facemask 5 week Use in Class III Malocclusion

SUMMARY:
Diverse viewpoints exist regarding the correlation between the conventional rapid maxillary expansion (RME) and facemask approach and the alternative RME and facemask hybrid technique (Alt-RAMEC) in terms of the degree of maxillary protraction. The findings of the study may offer a novel approach to protocol selection based on the anomaly's degree of severity. The objective of this investigation is to assess and contrast the skeletal and dentoalveolar outcomes of three distinct Alt-RAMEC techniques.

DETAILED DESCRIPTION:
Alternating rapid maxillary expansion and constriction (Alt-RAMEC) procedure is one of the most frequently used methods in the treatment of Class III cases caused by maxillary retrognathia. The objective of this investigation is to conduct a comparative analysis of the skeletal and dentofacial outcomes of three distinct techniques for maxillary protraction Following the primary recording, the patients were evaluated using bonded-type rapid maxillary expansion (RME) devices and three discrete Alt-RAMEC techniques (1, 3, and 5 weeks). Lateral cephalograms were obtained from a sample of 40 patients (18 males and 22 females) with a mean age of 10.64 ± 0.98. These images were taken both before (T1) and after the 6th month of facemask treatment (T2), and were subjected to total and local superimpositions. The Wilcoxon Sign, Kruskal-Wallis and Mann-Whitney U tests were used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary retrognathia (SNA ≤ 79°)
* Skeletal Class III malocclusion (ANB ≤ -1°)
* Anterior cross-bite
* Class III molar relationship
* Horizontal growth pattern (SN/Go-Gn < 30°)

Exclusion Criteria:

* Previous orthodontic treatment
* Systemic disorders

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-01-13 (Actual); Primary Completion 2012-07-15 (Actual); Study Completion 2012-08-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of Skeletal, Dental, and Soft Tissue Angular Measurements | 6 months
  Changes at the maxillary advancement, teeth positions and soft tissues amount were assessed in angular level.
  Skeletal measurements:
  Angular measurements: SNA (°), SNB (°), SN/S-Gn (Y-axis)(°), SN/Go-Gn (°), Ar-Go-Gn (°), SN/Go-Ar (°), and ANB (°) were measured.
  Dental measurements:
  Angular measurements: U1 to MaxP (°) for maxillary dentoalveolar measurements; L1-MandP (°) for mandibular dentoalveolar measurements; U1-L1 (°) for interdental measurements were performed.
  Soft tissue measurements: Changes at the upper and lower lip assessed.
  Angular measurements: G-Sn-Pg' (°), Nasolabial angle (°), and Labiomental angle (°) were measured.

SECONDARY OUTCOMES:
Evaluation of Skeletal, Dental, and Soft Tissue Millimetrical Measurements | 6 months
  Changes at the maxillary advancement, teeth positions and soft tissues amount were assessed in millimetrical level.
  Skeletal measurements:
  Millimetrical measurements: Co-A (mm) for maxillary skeletal measurement, Co-B (mm) for mandibular skeletal measurement, N-Me (mm), N-ANS (mm), and ANS-Me (mm) for maxillomandibular skeletal measurements were performed.
  Dental measurements:
  Millimetrical measurements: U1-MaxP (mm), U1-MaxVP (mm), U6-MaxP (mm), U6-MaxVP (mm) for maxillary dentoalveolar measurements; L1-MandP (mm), L1-MandVP (mm), L6-MandP (mm), L6-MandVP (mm) for mandibular dentoalveolar measurements; Overbite (mm) and overjet (mm) for interdental measurements were performed.
  Soft tissue measurements: Changes at the upper and lower lip assessed.
  Millimetrical measurements: Ls-S (mm) and Li-S (mm) were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Yılmaz Öğütlü, Dr., Study Director — Istanbul University; Gülsün Külekçi Çakan, Principal Investigator — Private Practitioner; Hülya Kılıçoğlu, Prof. Dr., Study Chair — Istanbul University; Hande Uzunçıbuk, Dr., Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No